CLINICAL TRIAL: NCT02859493
Title: Evaluation of the Effect of Saccharomyces Cerevisiae on the Improvement of the Conventional Treatment for Vulvo-vaginal Infection to Candida Spp (Local Administration)
Brief Title: Effect of Saccharomyces Cerevisiae on Vulvo-vaginal Candidiasis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: Lesaffre International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 15E2899
Record Dates: First submitted 2016-08-04; First posted 2016-08-09 (Estimated); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: Candidiasis, Vulvovaginal
MeSH Terms: conditions — Candidiasis, Vulvovaginal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saccharomyces cerevisiae (Active Comparator): Inactivated whole yeast Saccharomyces cerevisiae presented in vaginal capsules. 1 capsule a day for 14 days.
  Interventions: Device: Saccharomyces cerevisiae
- Maize starch and magnesium stearate (Placebo Comparator): Placebo presented in a vaginal capsule. 1 capsule a day for 14 days
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Saccharomyces cerevisiae
  Arms: Saccharomyces cerevisiae
Device: Placebo
  Arms: Maize starch and magnesium stearate

SUMMARY:
This study aims to evaluate the effect of a specific strain of Saccharomyces cerevisiae on improving the effectiveness of conventional treatment of vulvo-vaginal candidiasis. This is a randomized, double-blind, placebo-controlled study. The administration of yeast will be local (vaginal).

ELIGIBILITY:
Inclusion Criteria:

* Subject suffering from a vulvo-vaginal candidiasis (according to clinical examination) characterized by a vaginal discharge associated with any of the following symptoms: itching and burning vaginal feeling, dyspareunia and dysuria.
* Amenorrheic subject, or subject having a regular menstrual cycle.
* Subject psychologically able to understand the study related information and to give a written informed consent.
* Subject having given freely and expressly her informed consent.
* Subject able to comply with protocol requirements, as defined in the protocol.
* Subject affiliated to a health social security system.
* Female subjects of childbearing potential should use a medically accepted contraceptive regimen (except latex condom, latex diaphragm, spermicidal) during the D0-D14 period, since at least 12 weeks before the beginning of the study, during all the study and at least 1 month after the study end, at the investigator's discretion

Exclusion Criteria:

In terms of population

* Pregnant or nursing woman or planning a pregnancy during the study.
* Post-menopausal women.
* Subject who will have her period between the first and the second visit to the gynaecologist (between D0 and D7).
* Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship.
* Subject in a social or sanitary establishment.
* Subject suspected to be non-compliant according to the investigator's judgment.
* Subject enrolled in another clinical trial on the same test zone within the four previous weeks and during the study period, being in an exclusion period for a previous study, having tested a food supplement or a medication in the 4 previous weeks.
* Subject in an emergency situation. In terms of associated pathology
* Subject with a condition or receiving a medication which, in the investigator's judgment, put the subject at undue risk.
* Subject suffering from systemic diseases using concurrent therapy that may interfere with the evaluation of the study results.
* Subject with a known allergy to one of the component of the study products or to the medication (vaginal ovule and/or antifungal cream).
* Subject presenting an hypersensitivity to any antifungal of imidazole family or to one of the excipient.
* Uterine or vaginal bleeding of unknown origin
* Subject with known sexually transmitted infections such as Neisseria gonorrhoea, Chlamydia trachomatis, Treponema pallidum, herpes simplex, Trichomonas vaginalis, human papilloma virus or HIV 1 or 2.
* Immunocompromised subjects

Relating to previous or ongoing treatment

• Subject undergoing a topical treatment on the test area or a systemic or intravaginal treatment:

* antibiotics currently or within the past 2 weeks (systemic antibiotic are accepted if the treatment was stopped until the day before the inclusion visit)
* anti-fungal agents currently or within the past 2 weeks,
* anticoagulant within the past 2 weeks and during the study,
* anti-inflammatory medication and/or anti-histamines during the previous 2 weeks and during the study,
* corticosteroids during the 2 previous weeks and during the study,
* retinoids and/or immunosuppressors during the 3 previous months and during the study,
* any medication stabilized for less than one month.

In terms of lifestyle

* Subject planning to change her usual hygiene habits and products during the study.
* Subjects not willing to stop taking probiotics dietary supplements and food products enriched with probiotics.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Diminution of the vaginal load in Candida spp (Candida albicans, Candida glabrata) in subjects presenting a vulvo-vaginal candidosis | after 7 days and 14 days of treatment
  valuation of the effect of vaginal administration of Saccharomyces cerevisiae on the vaginal load in Candida spp (Candida albicans, Candida glabrata) in subjects presenting a vulvo-vaginal candidosis, by counting Candida spp in vaginal samples, before treatment and after 7 days and 14 days of treatment, in addition to a conventional medical treatment and in comparison to the placebo product.

CONTACTS AND LOCATIONS:
Locations (1):
- Dermscan, Villeurbanne, France

IPD SHARING:
Plan to Share IPD: No